CLINICAL TRIAL: NCT03079362
Title: SDR Monitoring in Children With Cerebral Palsy - a Retrospective Cohort Study
Brief Title: SDR Monitoring in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: SDR
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children: Children who underwent selective dorsal rhizotomy (SDR) including intraoperative neuromonitoring (IOM)

SUMMARY:
The study evaluates the anatomical distribution of the assessed Electromyogram (EMG) responses ensuring after sensory nerve root stimulation and obtained IOM grading during selective dorsal rhizotomy (SDR) with regard to level and, side of the body and gender as well as pain management and outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children with spastic cerebral palsy undergoing selective dorsal rhizotomy surgery including intraoperative neuromonitoring

Exclusion Criteria:

* > 21 years

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female pediatric and adolescent patients undergoing SDR
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2007-01-15 (Actual); Primary Completion 2014-11-27 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
The frequency distribution pattern of the grading assessed by SDR monitoring Electromyogram (EMG) procedure | During the operation

SECONDARY OUTCOMES:
Intensive care unit length of stay | Participants will be followed for the duration of hospital stay, an expected average of 1 day
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Ready to discharge | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Measured Pads-Score
Duration of ventilation | Participants will be followed for the duration of intensive care unit stay, an expected average of 1 day
  Measured in days and hours
Pain | Up to 12 months
  Measured by scales
Organ complications | Up to 12 months
Adverse reactions of pain therapy | Up to 12 months
Therapy of adverse reactions of pain therapy | Up to 12 months
Infections | Up to 12 months
Delirium | Up to 12 months
  Measured by Nu-DESC
Routine laboratory | Up to 12 months
Pain therapy | Up to 12 months
Temperature | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Satisfaction with pain therapy | Up to 12 months
  Rating scale
Positional control of epiperidural catheter | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Reoperations | Up to 12 months
Gross motor function measure | Up to 12 months
Gait analysis instrumented three dimensional | Up to 12 months
Strength | Up to 12 months
Spasticity | Up to 12 months
Range of motion | Up to 12 months
Gait | Up to 12 months
Functions scores | Up to 12 months
Gross motor function classification system | Up to 12 months
Modified Ashworth Scale | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité University Medicine -Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolter S, Spies C, Martin JH, Schulz M, Sarpong-Bengelsdorf A, Unger J, Thomale UW, Michael T, Murphy JF, Haberl H. Frequency distribution in intraoperative stimulation-evoked EMG responses during selective dorsal rhizotomy in children with cerebral palsy-part 1: clinical setting and neurophysiological procedure. Childs Nerv Syst. 2020 Sep;36(9):1945-1954. doi: 10.1007/s00381-020-04734-z. Epub 2020 Jun 23. PMID 32577878